CLINICAL TRIAL: NCT04790721
Title: How Much Does Technology Addiction in Youth Affect Academic Achievement, Musculoskeletal System and Quality of Life?
Brief Title: Relationship Between Academic Achievement, Musculoskeletal System, Quality of Life and Technology Addiction
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Ünal, PhD, Pamukkale University
Other Study IDs: 10.09.2019 / 15
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Technology Addiction; Musculoskeletal System; Quality of Life; Youth
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The increasing use of technological devices such as mobile phones and computers has become indispensable elements of daily life. Especially students are one of the groups that use communication tools most with the developing technology. This study was conducted to investigate the effect of technology addiction on academic achievement, musculoskeletal system and quality of life in young people.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 20-30, using smartphones and/or computers were included in the study.

Exclusion Criteria:

* Individuals who did not meet the inclusion criteria and had a physical-psycho-social condition that could affect the study were excluded from the study.

Ages: 20 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Our study is important in terms of determining the effects of not only smartphone use but also computer use addiction on health. For this reason, our study was conducted to investigate the effect of technology addiction on academic achievement, musculoskeletal system and quality of life on behalf of young people.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction Scale-Short Form | 5 minutes
  It is a 10-item scale assessed with a six-point Likert rating developed by Kwon et al. to measure the risk of smartphone addiction in adolescents.
Young Internet Addiction Test Short Form | 5 minutes
  Developed by Young and converted into short form by Pawlikowski et al., IAT-SF consists of 12 items (13,14). IAT-SF, for which Turkish validity and reliability study has also been carried out, is a five-point Likert (1 = Never, 5 = Very often) type scale. High scores on the scale indicate a high level of internet addiction
Cornell Musculoskeletal Discomfort Questionnaire | 5 minutes
  The survey indicates whether the pain or discomfort has affected the frequency of 11 different body regions (neck, shoulder, back, upper arm, waist, forearm, hip, upper leg, knee and lower leg) in the last 7 days, the severity of this situation and the ability to work. evaluates.
Short Form-36 | 5 minutes
  SF-36 Quality of life questionnaire was used as the general health questionnaire. SF-36, for which Turkish validity-reliability study was conducted, consists of eight subsections (general health perception, physical function, physical role limitation, emotional role limitation, social function, pain, energy, mental health) each varying between 2-10 questions.
Meaning of Life Questionnaire | 2 minutes
  Each item is evaluated according to a 7-graded response system (1: Strongly Disagree, 7: Strongly Agree). It is stated that as the score obtained from the questionnaire increases, life satisfaction increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)